CLINICAL TRIAL: NCT02799134
Title: Neural Mechanism of Cortisol Awakening Response Suppression Effect on Human High-order and Social Cognitions
Acronym: NMCARSEHHSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: qinshaozheng (Other)
Collaborators: Chinese Academy of Sciences (Other Government); Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, qinshaozheng, Professor, Beijing Normal University
Organization: Beijing Normal University (Other)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: ICBIR_A_0098_002
Record Dates: First submitted 2016-04-06; First posted 2016-06-14 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Healthy
Keywords: Cortisol Awakening Response suppression; Dexamethasone Suppression Test; high-order cognition; social cognition
MeSH Terms: interventions — Dexamethasone; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- group1 (Experimental): take Dexamethasone at 22:00 on the first day, 0.5mg
  Interventions: Drug: Dexamethasone
- group2 (Placebo Comparator): take Vitamin C at 22:00 on the first day, 0.5mg
  Interventions: Drug: Vitamin C
- group3 (Other): take Dexamethasone at 15:00 on the second day, 0.5mg
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone
  Arms: group1; group3
Drug: Vitamin C
  Arms: group2

SUMMARY:
CAR is short for cortisol awakening response. The neural mechanism of CAR effect on high-order cognition and social cognition is less known...

ELIGIBILITY:
Inclusion Criteria:

* Healthy college students.

Exclusion Criteria:

* Current or history of psychiatric or neurological illness.
* Current use of any medications.

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Cortisol Awakening Response Level(nmol/L) after Taking Dexamethasone | one year
  The dosage of Dexamethasone is 0.5mg.

CONTACTS AND LOCATIONS:
Overall Officials: Shaozheng Qin, Doctor, Study Chair — Beijing Normal University
Locations (1):
- Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided